CLINICAL TRIAL: NCT04360408
Title: The Energy Conservation Education Intervention For People With End-stage Kidney Disease Receiving Haemodialysis (EVEREST)
Brief Title: The Energy Conservation Education Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queensland University of Technology (Other)
Responsible Party: Principal Investigator, Sita Sharma, Principle Investigator, Queensland University of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSharma
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Fatigue; End Stage Kidney Disease; Quality of Life
Keywords: End-stage kidney disease, fatigue, haemodialysis, quality of life
MeSH Terms: conditions — Fatigue; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participant of the cluster randomised to the intervention group will receive both the usual care from their healthcare providers and EVEREST delivered by the researcher who is a nurse.
  Interventions: Other: Energy conservation education intervention for people with end-stage kidney disease receiving hemodialysis
- Control (No Intervention): Participants of the cluster randomised to the control group will receive usual care (standard care with no formalised, structured or tailored interventional to reduce symptom/s) from their healthcare providers

INTERVENTIONS:
Other: Energy conservation education intervention for people with end-stage kidney disease receiving hemodialysis — The total program consisting of three educational sessions (at Week -1, week -3 and week -5) and one booster session (week -10) over a period of 12 weeks. Participants will receive individual, face to face education during their regular HD session. Education will be provided over 30-45 minutes for the first session, 30 minutes in the next two sessions and 30-45 minutes for the booster session. The lead researcher, who is a nurse, will deliver the entire intervention to avoid information bias. The simple language will be used, and emphasis will be given on the objectives of each session.
  Arms: Intervention

SUMMARY:
Fatigue is the most common symptom reported by 70 - 85 % of people with end-stage kidney disease (ESKD) receiving haemodialysis (HD). Educational interventions involving energy conservation strategies are helpful in reducing fatigue. However, the effectiveness of energy conservation has not been previously studied in people with ESKD receiving HD. This study aims to develop and evaluate the effectiveness of energy conservation education intervention for people with end-stage kidney disease receiving haemodialysis (EVEREST) in Nepal.

Symptom Management Theory (SMT) will guide this study. A pragmatic cluster randomised controlled trial (pCRT) will be conducted in one dialysis centre in Nepal. People on HD who meet the eligibility criteria will be invited to participate. The primary outcome is fatigue severity and the secondary outcome are other renal symptoms, occupational performance and health-related quality of life. Intention to treat analysis will occur and will include a change in the primary and secondary outcome. The study will provide evidence about the feasibility and effectiveness of EVEREST for symptom management.

ELIGIBILITY:
Inclusion Criteria:

Participants diagnosed with ESKD and undergoing haemodialysis for ≥ 3 months, aged 18 years and above, able to speak and understand Nepali language and willing to participate will be included in this study.

Exclusion Criteria:

Participants who are in the early stage of CKD or not dependent on HD, those acutely ill, diagnosed with cognitive impairment and those who are not willing to participate will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Changes in Fatigue Symptom Inventory (FSI) | Baseline and week 4
  Fatigue Symptom Inventory (FSI) will be used to assess the severity, frequency, interference associated with fatigue and daily pattern of fatigue. The scale consists of 14 items rated on the 11-point items.
Changes in Fatigue Symptom Inventory (FSI) | Baseline and week 8
  The scale consists of 14 items rated on the 11-point items.
Changes in Fatigue Symptom Inventory (FSI) | Baseline and week 12
  The scale consists of 14 items rated on the 11-point items.

SECONDARY OUTCOMES:
Other renal symptoms | Baseline and Week 12
  Other renal symptoms will be measured using the renal version of the IPOS (IPOS-Renal). It is a short 11-item measure, combining the most common symptoms experienced by renal patients and additional items from IPOS on concerns beyond symptoms, such as information needs, practice issues, family anxiety during the past three days. Ten questions, including 23 subitems, covers physical and psychological symptoms, carer anxiety and practical issues with optional items for any other concern. Each item is scored using a five-point Likert scale for severity and total score reflect symptom burden.
Occupational Performance | Baseline and week 12
  The Canadian Occupational Performance Measure (COPM) is a valid and reliable instrument that measures the occupational performance. The COPM is designed to identify changes in the individual's personal perceptions of occupational performance over a period of time. Individual rates their performance within the area of self-care, productivity and leisure and satisfaction with their performance. Both scales range from 1-10, with higher values indicating better performance and greater satisfaction.
Health-related quality of life (HRQoL) | Baseline and Week 12
  Health-related quality of life will be measured using the SF-36 which is the 36-items self-administered survey of a patient's health. There are two distinct concepts measured by the SF-36 represented by the physical component summary (PCS) and mental component summary (MCS). For each sub-scale, items are scored using a Likert scale, summed and transformed on to a scale from 0 (worst health) to 100 (best health)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma S, Alexander KE, Green T, Wu ML, Bonner A. Energy conservation education intervention for people with end-stage kidney disease receiving haemodialysis (EVEREST): A two-arm parallel group study. Int J Nurs Stud. 2025 Jun;166:105032. doi: 10.1016/j.ijnurstu.2025.105032. Epub 2025 Feb 24. PMID 40101671
- [Derived] Sharma S, Alexander KE, Green T, Wu MW, Bonner A. Energy conservation education intervention for people with end-stage kidney disease receiving haemodialysis (EVEREST): protocol for a cluster randomised control trial. BMJ Open. 2022 Feb 21;12(2):e056544. doi: 10.1136/bmjopen-2021-056544. PMID 35190440